CLINICAL TRIAL: NCT01992276
Title: Multicenter, Randomized, Double-blind, Placebo-controlled Study to Evaluate the Effect of CR8020 and CR6261 in Hospitalized Patients With Influenza A Infection
Brief Title: Assessment of Efficacy of CR8020 and CR6261, Monoclonal Antibodies, Against Influenza Infection
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Due to preliminary efficacy results from an influenza challenge trial
Sponsor: Crucell Holland BV (Industry)
Collaborators: Division of Microbiology and Infectious Diseases (DMID) (Unknown); National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CR102576; 2013-003341-41 (EudraCT Number); CR6261CR8020FLZ2001 (Other: Crucell Holland BV)
Record Dates: First submitted 2013-11-11; First posted 2013-11-25 (Estimated); Last update posted 2014-03-04 (Estimated); Status verified 2014-03

CONDITIONS: Influenza
Keywords: Influenza; Virus; Monoclonal Antibody; Immunization; Treatment
MeSH Terms: conditions — Influenza, Human; Virus Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- CR8020 (Experimental): Investigational monoclonal antibody against influenza A viruses
  Interventions: Biological: CR8020
- CR6261 (Experimental): Investigational monoclonal antibody against influenza A viruses
  Interventions: Biological: CR6261
- Placebo (Placebo Comparator): Dextrose: 5% in water
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: CR8020 — 30 mg/kg administered as a single 2-hour intravenous infusion on Day 1
  Other Names: CR8020 30 mg/kg by iv infusion
  Arms: CR8020
Biological: CR6261 — 30 mg/kg administered as a single 2-hour intravenous infusion on Day 1
  Other Names: CR6261 30 mg/kg by iv infusion
  Arms: CR6261
Biological: Placebo — Administered as a single 2-hour intravenous infusion on Day 1
  Other Names: Placebo by iv infusion
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the rate of decline in quantitative viral load measured in hospitalized patients with Influenza A infection

DETAILED DESCRIPTION:
This is a randomized, placebo-controlled, double-blind phase IIa proof-of-concept study, designed to evaluate the effect of CR8020, CR6261, or placebo in hospitalized patients with influenza A infection that are receiving standard of care. Up to 262 participants will be randomized to receive 30 mg/kg of CR8020, 30 mg/kg of CR6261, or placebo. The study duration will be approximately 117 days for each participant. Prior to enrollment, participants will be screened to assess their eligibility. Eligible participants will be randomized to CR8020, CR6261, or placebo and study drug will be administered on Day 1. Participants will be followed up for 115 days in 9 visits on Days 2 to 8, Day 29, and Day 116 (end of study). After hospital discharge, the remaining follow-up visits will be performed as outpatient visits.

ELIGIBILITY:
Inclusion Criteria:

Participant requires hospitalization/ Each participant or his or her legally acceptable representative must sign an informed consent form/ Participant must be able to start the infusion within 36 hours from the time the screening specimen was collected/ A woman must either be not of childbearing potential or of childbearing potential and agrees to practice two forms of highly effective method of birth control/ A woman of childbearing potential must have a negative serum (beta human chorionic gonadotropin [beta hCG]) at screening/ A man who is sexually active with a woman of childbearing potential and has not had a vasectomy must agree to use a barrier method of birth control/

Exclusion Criteria:

Participant is a female who is pregnant or breastfeeding/ Participant undergoing peritoneal dialysis, hemodialysis or hemofiltration/ Participant has presence of any pre-existing illness that, in the opinion of the investigator, would place the participant at an unreasonably increased risk through participation in this study/ Participant has prior treatment with an experimental mAb; or receipt of IgG within 3 months or on chronic mAb treatment prior to enrollment/ Participant has known or suspected hypersensitivity to any of the CR8020 or CR6261 excipients (sucrose, L-histidine L-histidine monohydrochloride, polysorbate 20)/ Participant received an investigational product (including investigational vaccines) or used an investigational medical device within 60 days before the planned start of treatment, is currently enrolled in an interventional investigational study, or is an employee of the investigational site/

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-12; Primary Completion 2014-10 (Estimated); Study Completion 2015-02 (Estimated)

PRIMARY OUTCOMES:
Rate of decline in quantitative viral load | Baseline to Day 8

SECONDARY OUTCOMES:
Clinical improvement | Baseline to Day 15
  Daily influenza symptoms and signs:
  Four domains from the Influenza Intensity and Impact Questionnaire will be evaluated (scored 0-3: none, mild, moderate, severe):
  -Influenza symptoms (respiratory and systemic domains Impact on daily activities Impact on emotions Impact on others
Rate of decline in quantitative viral load (subjects not intubated at baseline) | Baseline to Day 8
Rate of decline in quantitative viral load (subjects intubated at baseline) | Baseline to Day 8
Rate of decline in quantitative viral load | Baseline to Day 8
Incidence of adverse events | Baseline to Day 116
Incidence of serious adverse events | Baseline to Day 116
Area under the curve of viral load | Baseline to Day 8
Clinical course for ICU patients | Baseline to Day 8
Length of hospital stay | The duration of hospital stay, an expected average of 7 days
Survival times | Baseline to Day 116
  Survival times measured from randomization to time of death

CONTACTS AND LOCATIONS:
Overall Officials: Crucell Holland BV Clinical Trial, Study Director — Crucell Holland BV
Locations (68):
- United States (21):
  - Fresno, California
  - Stanford, California
  - Washington D.C., District of Columbia
  - Tampa, Florida
  - Chicago, Illinois
  - Maywood, Illinois
  - Baltimore, Maryland
  - Detroit, Michigan
  - Royal Oak, Michigan
  - Troy, Michigan
  - Minneapolis, Minnesota
  - St Louis, Missouri
  - Hackensack, New Jersey
  - Somers Point, New Jersey
  - New York, New York
  - Rochester, New York
  - Winston-Salem, North Carolina
  - Dayton, Ohio
  - Wilkes-Barre, Pennsylvania
  - Nashville, Tennessee
  - Houston, Texas
- Australia (4):
  - Adelaide
  - Melbourne
  - Parkville - Vic
  - Westmead
- Belgium (4):
  - Brussels
  - Edegem
  - Ghent
  - Leuven
- Brazil (8):
  - Belo Horizonte
  - Campinas
  - Curitiba
  - Passo Fundo
  - Porto Alegre
  - Ribeirão Preto
  - São José do Rio Preto
  - São Paulo
- Sofia, Bulgaria
- Canada (2):
  - Toronto, Ontario
  - Toronto
- France (6):
  - Clermont-Ferrand
  - Limoges
  - Lyon
  - Paris
  - Rennes
  - Saint-Priest-en-Jarez
- Germany (4):
  - Donaustauf
  - Jena
  - Leipzig
  - Potsdam
- Netherlands (4):
  - Amsterdam
  - Apeldoorn
  - Leiden
  - Utrecht
- South Africa (3):
  - Benoni
  - Durban
  - Pretoria Gauteng
- Spain (8):
  - Alicante
  - Barcelona
  - Córdoba
  - Donostia / San Sebastian
  - Elche
  - Madrid
  - Santander
  - Tarragona
- Sweden (3):
  - Malmo
  - Stockholm
  - Uppsala